CLINICAL TRIAL: NCT02843542
Title: Localization of Parathyroid Adenoma by Fluorocholine Positron Emission Tomography/MRI (PET/MRI): A Prospective Pilot Study
Brief Title: Localization of Parathyroid Adenoma by Fluorocholine PET/MRI (Positron Emission Tomography -MRI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Avi Hefetz, MD, Assuta Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0012-16-ASMC
Record Dates: First submitted 2016-07-14; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Primary Hyperthyroidism
Keywords: Positron emission tomography-magnetic resonance imaging (PET-MR); Hyperthyroidism; Positron emission tomography-computed tomography (PET-CT)
MeSH Terms: conditions — Hyperthyroidism | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Other): primary hyperthyroidism patients that will be refered to the routine exams (PET-CT)
  Interventions: Device: PET-CT
- Study group (Other): primary hyperthyroidism patients that will be refered to the routine exams (PET-CT) and in addition will also undergo the PET-MR
  Interventions: Device: PET-MR; Device: PET-CT

INTERVENTIONS:
Device: PET-MR — Patients with Hyperthyroidism and surgery indication will be recruited and directed to imagine exams. In addition to the conservative 99mTc-MIBI and US, patients will also undergo 18FCH PET/MRI for detecting adenomas and their location.
  Arms: Study group
Device: PET-CT — Patients with Hyperthyroidism and surgery indication will be recruited and directed to imagine exams. In addition to the conservative 99mTc-MIBI and US, patients will also undergo PET-CT for detecting adenomas and their location.

SUMMARY:
A comparative prospective study to evaluate different imaging modalities (pet-ct and pet-mr) prior to surgery in parathyroid tumor patients.

DETAILED DESCRIPTION:
Patients with Hyperthyroidism and surgery indication will be recruited and directed to imagine exams. in addition to the conservative 99mTc-MIBI (methoxyisobutylisonitrile) and US, patients will also undergo 18FCH (¹⁸F-choline) PET/MRI for detecting adenomas and their location. imaging experts will decode the imaging exams. sensitivity and specificity of the exams will be examined.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the criteria accepted in the World Health Organization (WHO) analysis:

* Symptomatic patients (constipation, depression, peptic ulcer, pathologic fractures, chronic fatigue, pain from a urinary tract stones etc..)

or at least one of the following criteria:

* Blood calcium levels above 1 more than normal
* Creatinine clearance decreased in 30% from age expected
* Urine Creatinine above 400 mg in 24 hours

Exclusion Criteria:

* Patients with hyperthyroidism secondary and tertiary (secondary to kidney disease)
* Patients who are not eligible to sign an informed consent
* Pregnant women
* Patients with sensitivity (allergy) technetium or 18FCH

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Adenomas size and location | 24 months
  Location of adenomas by a report analyzing the pathological examination (PET-CT/PET-MR output).

SECONDARY OUTCOMES:
Parathyroid hormone levels | 24 months
  approval late addition level of parathyroid hormone (PTH) before and during the course of the operation after the conclusion of adenomas (Hormone levels).
Chronic disease duration | 24 months
  time from chronic diseases indication and duration of symptoms measured in months (from the medical records).
Disease related medication consumption | 24 months
  Disease related medication consumption measured in miligram (mg) for each medication (from medical records).

CONTACTS AND LOCATIONS:
Overall Officials: Avi hefetz, MD, Principal Investigator — Assuta Medical Center
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No